CLINICAL TRIAL: NCT02144298
Title: The Perioperative Course of Sublingual Microcirculatory Alterations in Patients Undergoing Extracorporeal Flow Conditions: Cold Blood Compared With Cristalloid Cardioplegia
Brief Title: The Sublingual Microcirculatory Alterations in Patients Undergoing Extracorporeal Flow Conditions
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Matty Koopmans, MSc, Frisius Medisch Centrum
Other Study IDs: ATADEK 2013-540
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Microcirculatory Alterations
Keywords: microcirculation; coronary artery bypass grafting; cold blood cardioplegia; cristalloid cardioplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cold blood cardioplegia: observe the perioperative course of sublingual microcirculatory alterations in patients undergoing coronary artery bypass grafting (CABG) using cold blood cardioplegia.
- cristalloid cardioplegia: observe the perioperative course of sublingual microcirculatory alterations in patients undergoing coronary artery bypass grafting (CABG) using cristalloid cardioplegia.

SUMMARY:
The aim of this study is to observe the perioperative course of sublingual microcirculatory alterations in patients undergoing coronary artery bypass grafting (CABG) using cold blood compared with cristalloid cardioplegia. Additionally the impact of changes in hemodynamic parameters, blood gas, laboratory findings and standart therapy for intra and early postoperative period was studied. Intubation time, ICU stay, hospital stay, ICU readmission, morbidity and mortality were recorded.

DETAILED DESCRIPTION:
The microcirculatory measurements were obtained in both groups in the sublingual mucosa using Cytocam imaging. The probe was handheld. Different precautions were taken and steps followed to obtain images of adequate quality and to ensure good reproducibility.

Images were made after induction of anesthesia (t0), before CBP 5 minutes after heparine (t1), 5 minutes after CBP beginning (t2), during CBP 10 minutes after crossclamp beginning (t3), after crossclamp ending when heart begins to beat (t4), after CBP 10 minutes after protamine (t5).

Additional images were made before (tc0) and after (tc1) vasoactive medication; before (tv0) and after (tv1) volume administration; before (tb0) and after (tb1) blood administration, (FFP, PLT).

At each timepoint adequate focus depth and contrast were noticed. Three steady images of 6 seconds were acquired and recorded on a device controller based on a powerful medical grade computer which is used for image storage and analysis.

Additionally macrocirculatory measurements were obtained at the same timepoints. Hemodynamic variables, temperature, blood gas, INVOS, StO2, laboratory findings and standart therapy were recorded. Additionally intubation time, ICU stay, hospital stay, ICU readmission, morbidity and mortality were studied.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing coronary artery bypass grafting (CABG)

Exclusion Criteria:

* previous heart and oral surgery
* age below 18 years,
* emergency surgery
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: of patients undergoing coronary artery bypass grafting (CABG) using cristalloid (n=10) or cold blood (n=10) cardioplegia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
functional capillary density | moment of measurement
  functional capillary density is expected to be lower in the cryaloide group

SECONDARY OUTCOMES:
percentage perfused density | time of measurement
  a higher percentage of perfused vessel density is expected in the blood group

CONTACTS AND LOCATIONS:
Overall Officials: Can Ince, Prof, Principal Investigator — Medical Centre Amsterdam
Locations (1):
- Acıbadem University Hospital, Istanbul, Turkey (Türkiye)